CLINICAL TRIAL: NCT06985186
Title: The Effect of Adenomyosis Following Ultra-long GnRH Agonists With or Without Aromatase Inhibitors on ART Outcomes (AURA Trial): a Randomized Controlled Trial
Brief Title: Does The Addition Of Letrozole To Ultra-Long GnRH Agonists Help Adenomyosis Patients in ART? The AURA Trial
Acronym: AURA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AURA Trial
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Adenomyosis of Uterus; Infertility Assisted Reproductive Technology
Keywords: adenomyosis; infertility; Ultra-Long GnRH Agonists; Aromatase inhibitor; IVF outcomes; assisted reproductive technology; egg-donation
MeSH Terms: conditions — Adenomyosis; Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultra-Long GnRH Agonists (Active Comparator): All patients will receive a depot injection of the long-acting GnRH agonist, intramuscularly, once (11.25mg) or every 28 days (3.75mg) for at least 3 months prior to embryo transfer. The first injection of GnRH agonist will be administered during the menstrual phase of the cycle.
  Interventions: Drug: Ultra-Long GnRH Agonists
- Ultra-Long GnRH Agonists + Letrozole (Experimental): All patients will receive a depot injection of the long-acting GnRH agonist, intramuscularly, once (11.25mg) or every 28 days (3.75mg) for at least 3 months prior to embryo transfer. Upon initiation of the GnRH agonist, patients will also receive 2.5mg of Letrozole every 12h for 60 days. The start of therapy will be during the menstrual phase of the cycle.
  Interventions: Drug: Ultra-Long GnRH Agonists + Letrozole

INTERVENTIONS:
Drug: Ultra-Long GnRH Agonists + Letrozole — All patients will receive a depot injection of the long-acting GnRH agonist, intramuscularly, once (11.25mg) or every 28 days (3.75mg) for at least 3 months prior to embryo transfer. Upon initiation of the GnRH agonist, patients will also receive 2.5mg of Letrozole every 12h for 60 days. The start of therapy will be during the menstrual phase of the cycle.
  Arms: Ultra-Long GnRH Agonists + Letrozole
Drug: Ultra-Long GnRH Agonists — All patients will receive a depot injection of the long-acting GnRH agonist, intramuscularly, once (11.25mg) or every 28 days (3.75mg) for at least 3 months prior to embryo transfer. The first injection of GnRH agonist will be administered during the menstrual phase of the cycle.
  Arms: Ultra-Long GnRH Agonists

SUMMARY:
The AURA Trial seeks to improve fertility treatment for women affected by a condition known as adenomyosis. Adenomyosis often leads to heavy menstrual bleeding, pelvic pain, dyspareunia and can make it more difficult to achieve and maintain a healthy pregnancy.

In this randomized controlled trial participating women ≥ 18 years of age with a confirmed imaging diagnosis of adenomyosis according to Morphological Uterus Sonographic Assessment (MUSA) consensus will first undergo a thorough assessment. This initial workup includes reviewing medical history, assessing the characteristics of the uterus (volume, myometrial architecture, shape of the uterine cavity, stiffness, etc.) via 2D/3D transvaginal ultrasound, and obtaining blood tests to establish baseline hormone levels.

Once enrolled, each participant will be assigned at random-without prior knowledge by either the woman or her care team-to one of two 90-day pre-treatment regimens. The first group will receive monthly injections of a GnRH agonist, a medication that temporarily suppresses ovarian function and lowers estrogen levels. The second group will follow the same injection schedule but will also take daily letrozole tablets, an aromatase inhibitor that further reduces estrogen production. The hope is that this combined approach will calm the inflammatory environment caused by adenomyosis, promote a more receptive uterus, and ultimately increase the likelihood of an embryo developing beyond the critical 12-week mark.

At the end of the 90-day protocol, and after repeating all evaluations carried out during the enrolment phase, all women will proceed with the planned assisted reproductive technology cycle with the usual careful monitoring until the day of emrbyo transfer. To ensure correct interpretation of the results and to minimise the potential effect of any incompetent oocytes, only euploid embryos evaluated by pre-implantation genetic test or embryos derived from donated oocytes will be transferred. Pregnancy will be assessed first with a blood test, followed by an ultrasound scan at approximately six or seven weeks to confirm a clinical pregnancy. An ongoing pregnancy, defined by the detection of the fetal heartbeat beyond the 12th week, is the main measure of success.

By participating in AURA, women and their families not only gain access to cutting-edge clinical care but also contribute valuable knowledge that could shape future standard treatments for adenomyosis-related infertility. For further information or to explore participation, please reach out to the Instituto Bernebu Assisted Reproduction Center, where our team is ready to guide you through every step of this important study.

ELIGIBILITY:
Inclusion Criteria:

- Infertile patients affected by adenomyosis diagnosed by 2D-3D transvaginal ultrasound according to revised Morphological Uterus Sonographic Assessment consensus.

Exclusion Criteria:

* concomitant uterine fibroids,
* Müllerian malformations,
* endometrial pathology,
* thin endometrium,
* hydrosalpinx,
* mucometra,
* previous surgery except for previous cesarean section,
* coagulation disorders,
* untreated endocrinopathies,
* severe seminal pathologies,
* double ET,
* ET different from the first one after adenomyosis treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer
  An ongoing pregnancy was defined as each pregnancy showing a positive heartbeat at ultrasound after 12 weeks of gestation

SECONDARY OUTCOMES:
Implantation rate | 6 to 7 weeks after transfer
  The number of gestational sacs observed divided by the number of embryos transferred
Miscarriage rate | 22 weeks after embryo transfer
  The spontaneous loss of two or more clinical pregnancies prior to 22 completed weeks of gestational age

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes